CLINICAL TRIAL: NCT03765749
Title: Empirical Antibiotic and Outcome in Community-onset Bacteremia Caused by Third Generation Cephalosporin Resistant Enterobacteriaceae
Brief Title: Empirical Antibiotic and Outcome in Community-onset Bacteremia
Status: Completed | Type: Observational
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Principal Investigator, Vasin Vasikasin, Principal Investigator, Phramongkutklao College of Medicine and Hospital
Other Study IDs: PMK-032
Record Dates: First submitted 2018-03-22; First posted 2018-12-05 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Community onset 3rd generation cephalosporin resistant entero: Patient with Community onset third generation cephalosporin resistant enterobacteriaceae bacteremia who received inappropriate Antibiotic
- Nosocomial onset 3rd generation cephalosporin resistant ente: Patient with Nosocomial onset third generation cephalosporin resistant enterobacteriaceae bacteremia who received appropriate Antibiotic

SUMMARY:
Empirical antibiotic and outcome in Community-onset Bacteremia Caused by third generation cephalosporin resistant Enterobacteriaceae

DETAILED DESCRIPTION:
Prospective cohort study is conducted for monitoring outcomes and risk factors among community-onset bacteremia caused by third generation cephalosporin resistant enterobacteriaceae.

Primary endpoint is mortality rate among those who received initially inappropriate antimicrobial which switch to appropriate antimicrobial later when culture and antimicrobial susceptibility test reported among community-onset bacteremia caused by third generation cephalosporin resistant enterobacteriaceae.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Community-onset Bacteremia Caused by third generation cephalosporin resistant Enterobacteriaceae. Age > 18 years

Exclusion Criteria:

* Pregnancy
* Polymicrobial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with community-onset bacteremia caused by third generation cephalosporin resistant enterobacteriaceae. Age > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate among community-onset bacteremia caused by third generation cephalosporin resistant enterobacteriaceae | January 2018 - march 2019

CONTACTS AND LOCATIONS:
Locations (1):
- Worapong Nasomsong, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nasomsong W, Changpradub D, Vasikasin V. Impact of Inappropriate Empirical Antibiotic on Outcomes in Community-acquired Third Generation Cephalosporin Resistant Enterobacterales Bacteremia. Infect Chemother. 2022 Dec;54(4):722-732. doi: 10.3947/ic.2022.0096. PMID 36596682